CLINICAL TRIAL: NCT06789757
Title: An Open Label Phase II Study of Atezolizumab, Bevacizumab and Memantine in Patients With Hepatocellular Carcinoma
Brief Title: The Study of Atezolizumab, Bevacizumab and Memantine in Patients With Hepatocellular Carcinoma (HCC)
Acronym: (HCC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INOVA-2023-74
Record Dates: First submitted 2024-11-13; First posted 2025-01-23 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Atezolizumab; Bevacizumab; Memantine
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Memantine; Bevacizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Addition of Memantine to Atezolizumab and Bevacizumab (the current systemic standard of care) (Experimental): The study intervention consists of the use of the triplet therapy (atezolizumab, bevacizumab, and memantine) given in 21-day cycles over six months.
  Interventions: Drug: Memantine Hydrochloride; Drug: Bevacizumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Memantine Hydrochloride — Memantine (5mg) is an N-methyl-D-aspartate (NMDA) receptor antagonist given in 21-day cycles over six months in combination with Bevacizumab and Atezolizumab. Each week memantine will be escalated by 5mg as tolerated
  Other Names: Namenda
Drug: Bevacizumab — Bevacizumab (15mg/kg) is a vascular endothelial growth factor inhibitor given in 21-day cycles over six months in combination with Memantine and Atezolizumab.
  Other Names: Avastin
Drug: Atezolizumab — Atezolizumab (1200mg) is a programmed death-ligand 1 (PD-L1) blocking antibody given in 21-day cycles over six months in combination with Memantine and Bevacizumab
  Other Names: Tecentriq

SUMMARY:
The purpose of this research is to see the effect of triplet therapy with atezolizumab, bevacizumab, and memantine in treatment of your hepatocellular carcinoma.

DETAILED DESCRIPTION:
The goal of this study is to investigate the impact of targeting the NMDA receptor pathway, by enrolling patients with hepatocellular carcinoma undergoing systemic therapy. The study will involve adding memantine to the standard treatment of atezolizumab and bevacizumab, administered in 21-day cycles over six months. Patients will complete quality of life surveys at each cycle to assess their well-being and cancer-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Patients have newly diagnosed and previously untreated, histologically or radiologically confirmed hepatocellular carcinoma with at least one lesion that is measurable by RECIST 1.1 criteria. A prior HCC lesion that was treated surgically or by radiation is allowed as long as it was at least 2 years or more from the current HCC diagnosis.
3. Patient's cancer must be deemed locally advanced and unresectable
4. Patients must have a Childs-Pugh cirrhosis score of A5 or A6.
5. Eastern Cooperative Oncology Group Performance Status of 0-1.
6. Patients must have bone marrow and organ function as defined below:

   * Absolute Neutrophil Count ≥ 1,500/μL
   * Platelets ≥ 100,000/μL
   * Hemoglobin ≥ 90 g/L (9g/dL)
   * Total Bilirubin ≤ 3 x ULN
   * AST(SGOT)/ALT(SGPT)/Alkaline Phosphatase ≤ 3 x ULN Or ≤5x ULN if due to liver involvement by tumor
   * Creatinine ≤ 2.0 mg/dL
   * eGFR (using Cockcroft Gault equation) > 40ml/min
7. Chemotherapy is harmful to the human fetus. For this reason, sexually active males and females with partners of childbearing potential must agree to use an accepted and effective method of contraception prior to study entry and for the duration of the study.
8. Patients must demonstrate the ability to understand and the willingness to sign a written informed consent document.
9. Men and women, regardless of race, ethnic group, or sexual orientation are eligible for this study.
10. Patient must be able to swallow oral medication.

Exclusion Criteria:

1. Patients with Childs-Pugh B or C cirrhosis.
2. Female patients who are pregnant or breast-feeding.
3. Concomitant illness that would prevent adequate patient assessment or in the investigators' opinion pose an added risk for study participants.
4. Any history or evidence of severe illness or any other condition that would make the patient, in the opinion of the investigator unsuitable for the study. This would include any uncontrolled or untreated viral infection such as HIV, HBV, HCV etc.
5. Subject is enrolled in a separate interventional clinical trial.
6. Active tuberculosis.
7. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
8. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
9. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or bevacizumab formulation.
10. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
11. Uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at study entry.
12. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment.
13. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

18. Active, untreated grade 2 or 3 varices. Patients with treated varices to the point that they are grade 1 or less will be allowed.

19. Patients already on memantine for any reason prior to enrollment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2028-01-27 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of patients who are treated with the combination of atezolizumab, bevacizumab, and memantine. | Up to 2 years
  The effectiveness of the combination therapy using Azozolizumab, Bevacizumab,and Memantine in relation to the Objective Response Rate (ORR), defined as the proportion of complete or partial responses to the treatment by the response evaluation criteria for solid tumors(RECIST) 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Winer, MD, Principal Investigator — Principal Investigator
Locations (2):
- United States (2):
  - Inova Schar Cancer Institute - Fair Oaks, Fairfax, Virginia
  - Inova Health Care Service, Falls Church, Virginia

REFERENCES:
- [Background] Cabrera R, Nelson DR. Review article: the management of hepatocellular carcinoma. Aliment Pharmacol Ther. 2010 Feb 15;31(4):461-76. doi: 10.1111/j.1365-2036.2009.04200.x. Epub 2009 Nov 19. PMID 19925500
- [Background] Rawla P, Sunkara T, Muralidharan P, Raj JP. Update in global trends and aetiology of hepatocellular carcinoma. Contemp Oncol (Pozn). 2018;22(3):141-150. doi: 10.5114/wo.2018.78941. Epub 2018 Sep 30. PMID 30455585
- [Background] El-Serag HB, Kanwal F. Epidemiology of hepatocellular carcinoma in the United States: where are we? Where do we go? Hepatology. 2014 Nov;60(5):1767-75. doi: 10.1002/hep.27222. Epub 2014 Aug 25. No abstract available. PMID 24839253
- [Background] Liu P, Xie SH, Hu S, Cheng X, Gao T, Zhang C, Song Z. Age-specific sex difference in the incidence of hepatocellular carcinoma in the United States. Oncotarget. 2017 Jul 12;8(40):68131-68137. doi: 10.18632/oncotarget.19245. eCollection 2017 Sep 15. PMID 28978103
- [Background] Kim E, Viatour P. Hepatocellular carcinoma: old friends and new tricks. Exp Mol Med. 2020 Dec;52(12):1898-1907. doi: 10.1038/s12276-020-00527-1. Epub 2020 Dec 2. PMID 33268834
- [Background] Amit S, Jorge A M. Screening for hepatocellular carcinoma. Gastroenterol Hepatol (N Y). 2008 Mar;4(3):201-8. PMID 21904498
- [Background] Singal AG, Lampertico P, Nahon P. Epidemiology and surveillance for hepatocellular carcinoma: New trends. J Hepatol. 2020 Feb;72(2):250-261. doi: 10.1016/j.jhep.2019.08.025. PMID 31954490